CLINICAL TRIAL: NCT03315442
Title: Increased Static Postural Sway After Energy Drink Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Martin Rosario, Assistant Professor, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: A2540116
Record Dates: First submitted 2017-09-08; First posted 2017-10-20 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Disorder
Keywords: Fluid; Balance
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: 20 healthy adults, (11 males; 9 females) averaging 26.1 years of age, stood on a MatScan™ pressure mat, which measured center of pressure (CoP), anteroposterior (AP) and mediolateral (ML) postural sways during eight different balance tests (BALT's). BALT's were designed to alter or cancel the systems involved in postural control: visual, vestibular and somatosensory. Subjects were randomly assigned to a caffeine group and an energy drink group. MANOVA analysis was performed for all variables of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine Group (Sham Comparator): Caffeine group consumed 200mg of caffeine one time.
  Interventions: Other: Caffeine versus Energy Drink
- Energy Drink Group (Experimental): The energy drink group consumed 1 16 ounces energy drink one time.
  Interventions: Other: Caffeine versus Energy Drink

INTERVENTIONS:
Other: Caffeine versus Energy Drink — Caffeine group consumed 200mg of caffeine one time, while the energy drink group consumed 1 16 ounces of energy drink.

SUMMARY:
Background & Purpose: Energy drinks consumption continues to grow since its appearance in the United States in 1997. Available evidence indicates that caffeine, their main ingredient, can alter the central nervous system (CNS). However, it is unknown how energy drinks adjust the CNS postural control mechanism. The purpose of this study was to investigate how energy drinks can affect postural control after sensory perturbations during stance.

Methods: 20 healthy adults, (11 males; 9 females) averaging 26.1 years of age, stood on a pressure mat, which measured center of pressure (CoP), anteroposterior (AP) and mediolateral (ML) postural sways during eight different balance tests (BALT's). BALT's were designed to alter or cancel the systems involved in postural control: visual, vestibular and somatosensory. Subjects were randomly assigned to a caffeine group and an energy drink group. MANOVA analysis was performed for all variables of interest.

DETAILED DESCRIPTION:
Methods General Protocol

After signing the informed consent and reviewing the inclusion and exclusion criteria, participants were subjected to a preliminary screening of participation using a list of questions and the American college sports medicine Health / Fitness Facility Questionnaire. This questionnaire's purpose is to ensure the safety of the participants to engage in physical activity by assessing the subjects and family history of cardiovascular diseases. Afterwards, the Investigators assessed subjects' vital signs, blood pressure, pulse, and spO2, to ensure subjects were able to participate in physical activity safely ingest a moderate intake of caffeine without complications. Since postural control is negatively correlated with increased adiposity, weight and height data were measured to obtain a classification according to the Body Mass Index. A range of 18.5 to 29.9 was required to participate. During the physical examinations the subjects also performed a Romberg test to rule out any obvious impairment in static balance, a modified Sit and Reach Test for the evaluation of functional flexibility, Sit to Stand Test (30 Seconds) for the assessment of lower limb functional strength, and a Step Test to evaluate the response of the cardiovascular system to a submaximal cardio test. After the physical examination, the participants had a rest period between 10-20 minutes before starting the balance tests protocol of (BALT's).

Procedure

Each participant from both groups performed eight balance tests (BALT's) which alter or cancel, individually or combined, sensory input from the sensory systems involved in postural control. The order of the tests was changed systematically between subjects; therefore, they did not perform the tests in the same order to eliminate external factors such as fatigue or accommodation to the BALT's, which could alter the results. The BALT's were conducted on the (TekScan, Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose. The subjects stood for 30 seconds on the pressure platform during each test.

The first 4 BALT's were carried out by placing the pressure platform on the floor, a stable surface. These tests were: 1) Open Eyes (EO) with a fixed point to evaluate all the systems involved in the postural control (visual, vestibular, somatosensory); 2) Eyes Closed (EC) to evaluate the vestibular and somatosensory system, while eliminating the visual sensory input; 3) Eyes Open while actively moving the head up and down (HUD) to evaluate the visual and somatosensory system, while altering the vestibular system with head movements (EO HUD) (For HUD movements a metronome 2/4 60 BPM was used to maintain a fixed frequency of about one spin per second in motion); 4) Eyes closed and actively moving the head up and down (EC HUD) to assess the effect of removing the visual input, in combination of an alteration of the vestibular system with the head up and down movements.

The remaining 4 BALT's were the same as the four previously mentioned tests with the difference that the subject stood on an unstable surface (foam mat) that was placed on top of the pressure platform to alter the somatosensory (proprioceptive) system.

After the initial eight pre BALT's, to the experimental group, 160 mg of caffeine was given through one energy drink (16 ounces). Monster energy drink was chosen because, unlike other energy drink brands, the label of Monster Energy drink exhibits the guarana additive, a potential CNS stimulant, in its nutritional label. To the control group, Investigators gave a caffeine pill of 200mg, a moderate dose in healthy adults which has been used in numerous studies on different topics and has not been associated with adverse effects such as toxicity, cardiovascular effects, behavior changes, among other things. Because peak absorption of caffeine is reached within 30-45 minutes after the ingestion of caffeine/energy drink, there was a rest period of 30 minutes. Vital signs were measured after the rest period, for the third time. The same 8 BALT's were then performed, for post ingestion results.

ELIGIBILITY:
Inclusion Criteria:

* subjects between 21 to 40 years of age
* functional flexibility in the lower extremities
* functional muscular strength in the lower extremities
* completing the American College Sports Medicine Health/Fitness Facility Pre-participation screening Questionnaire
* Body Mass Index of 18.5 to 29.9
* arterial blood pressure less than or equal to 140/90 mmHg
* pulse at rest between 45-90 beats per minute (BPM) 95% or more of oxygen saturation (spO2).

Exclusion Criteria:

* subjects under the age of 21 and over the age of 40
* answering any questions affirmative on the pre-participation questionnaire
* cardiovascular problems
* severe balance problems
* taking any sedative or stimulant medications
* medical history of any neurological condition
* a fall in the last three months
* having undergone a surgical procedure in the past six months
* pain in the lower extremities and lower back
* have suffered a lower back injury and in the lower extremities in the last six months
* pregnant or suspecting pregnancy
* experienced adverse effects after caffeine consumption
* caffeine consumption 12 hours before the study intervention
* allergies to one of the energy drink ingredients, and 15) people unable to consent.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2017-01-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Center of Pressure and sway EYES OPEN | 30 minutes after caffeine or energy drink consumption
  Open Eyes (EO) with a fixed point to evaluate all the systems involved in the postural control. This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.
Center of Pressure and sway EYES CLOSED | 30 minutes after caffeine or energy drink consumption
  Eyes Closed (EC) to evaluate the vestibular and somatosensory system, while eliminating the visual sensory input. This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.
Center of Pressure and sway EYES HEAD UP AND DOWN | 30 minutes after caffeine or energy drink consumption
  Eyes Open while actively moving the head up and down (HUD) to evaluate the visual and somatosensory system, while altering the vestibular system with head movements (EO HUD) (For HUD movements a metronome 2/4 60 BPM was used to maintain a fixed frequency of about one spin per second in motion. This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.
Center of Pressure and sway CLOSED HEAD UP AND DOWN | 30 minutes after caffeine or energy drink consumption
  Eyes closed and actively moving the head up and down (EC HUD) to assess the effect of removing the visual input, in a combination of an alteration of the vestibular system with the head up and down movements. This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.
Center of Pressure and sway EYES OPEN ON FOAM | 30 minutes after caffeine or energy drink consumption
  standing on the unstable surface to evaluate the visual and vestibular system while the somatosensory is altered. This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.
Center of Pressure and sway EYES CLOSED ON FOAM | 30 minutes after caffeine or energy drink consumption
  Eyes Closed (MAT EO), standing on the unstable surface to evaluate the vestibular system (the somatosensory was modified and the visual system removed). This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.
Center of Pressure and sway EYES OPEN HEAD UP AND DOWN | 30 minutes after caffeine or energy drink consumption
  Eyes Open (MAT EO HUD) while actively moving the head up and down to evaluate the visual system, while altering the vestibular and somatosensory system. This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.
Center of Pressure and sway EYES CLOSED HEAD UP AND DOWN | 30 minutes after caffeine or energy drink consumption
  Eyes Closed (MAT EC HUD) while actively moving the head up and down (in this test all three systems were altered). The same frequency of motion used for BALT's 3 and 4 in the stable surface (one spin per second, 60 BPM) was maintained for the BALT's with HUD movements on the unstable surface. This study used (Boston, MA) a pressure platform containing sensors that measure a displacement of the center of pressure in centimeters squared (cm2) (CoP), anteroposterior (AP), and mediolateral (ML) sway in centimeters (cm). The data collected from the pressure mat was analyzed with Sway Analysis Module (SAM) software designed for this purpose.

SECONDARY OUTCOMES:
Body Mass Index | Pre Balance Test-Assessment
  kg/m^2
Weight | Pre Balance Test-Assessment
  kilograms
Height | Pre Balance Test-Assessment
  meters

CONTACTS AND LOCATIONS:
Locations (1):
- Biomechanics Laboratory of the Doctoral Program in Physical Therapy at the School of Health Professions in the Medical Sciences Campus, University of Puerto Rico (UPR-MSC)., San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No